CLINICAL TRIAL: NCT03031886
Title: Energy Flux and Fat Oxidation Using Low and High Glycaemic Index Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investogator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2015/01085
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes; Obesity; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State

STUDY DESIGN:
Intervention Model Description: A randomized,crossover design with either a low or high GI diet with a 5 day washout period in between the 2 interventions..
Who Masked: Participant, Investigator
Masking Description: Double blinded, subjects was blinded from knowing if foods were low or high GI, researchers analyzing the data were blinded from food preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high GI (Experimental): Cereal, milk, tea, cheese, steamed glutinous rice with chicken, carrots, bread, strawberry jam, margarine, high GI sweetener (sucrose).
  Interventions: Other: high glycaemic index intervention
- Low GI (Experimental): Cereal, milk, tea, steamed basmati rice with chicken, spinach, bread, strawberry jam, low GI sweetener (isomaltulose).
  Interventions: Other: low glycaemic index intervention

INTERVENTIONS:
Other: low glycaemic index intervention — Low GI sweetener would be added to the treatment meals. 30 grams of isomaltulose to dinner and breakfast and 20 grams of isomaltulose to lunch and snack.
  Arms: Low GI
Other: high glycaemic index intervention — High GI sweetener would be added to the treatment meals. 30 grams of sucrose to dinner and breakfast and 20 grams of sucrose to lunch and snack.
  Arms: high GI

SUMMARY:
Purpose: This study is carried out to determine the effect of GI on 24 hour blood glucose profiles and energy regulation in Asians when fed a normal diet modulated with sweeteners.

DETAILED DESCRIPTION:
The GI is a method of classifying foods based on the food's ability to raise the blood glucose level. Low GI foods are recommended as they have a lower impact on blood glucose concentrations. The research sets out to determine the effect of GI on 24 hour blood glucose profiles and energy regulation in Asians. Healthy, normal-weight and overweight, Chinese males will be recruited. There will be two sessions (consisting of three days for each session) where they will consume either a high or low glycaemic index dinner at home and a high or low GI breakfast, lunch and snack on the next day (in the whole body calorimeter). There will be at least five days in between the two sessions. Their glycaemic response will be measured using a Continuous Glucose Monitoring System (CGMS) throughout the period, while substrate oxidation will be measured over 10 hours in the calorimeter (from breakfast, lunch and snack). This study specifically attempts to see whether the inclusion of a low GI sweetener in a mixed meal sequence can impact blood glucose levels and energy regulation in Asians. The study is important in that it will enable us to compute the rate of fat oxidation and how it is influenced when subjects are fed a mixed meals modulated to be high GI (increased glucose excursions) or low GI (moderated glucose) over 24 hours in healthy Asians. Obesity and diabetes rates are increasing exponentially in Asian populations and Singapore is no exception. Devising ways and means to staunch the escalation is therefore a priority. The findings of the research will contribute towards the long-term objectives of developing dietary guidelines for weight and glycaemic control. The study data will also be important for the provision of practical food-based advocacy for better weight and glycaemic control in Asians.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, male
* Age between 21-40 years
* Body mass index between 17 to 28 kg/m2
* Normal blood pressure (<140/80 Hgmm)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Having any metabolic diseases (such as diabetes, hypertension etc)
* One prescription medication
* Partaking in sports at the competitive and/or endurance levels
* Allergic/intolerant to any of the test foods
* Intentionally restricting food intake
* Smoking

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — men only
Enrollment: 20 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | 3 hours post consumption
  The blood glucose response to low and high GI test foods measured 2 hours post consumption using the Continuous Glucose Monitoring System (CGMS)
Daily blood glucose profile | 24 hours
  The daily total blood glucose response is measured for each low and high GI treatment as the area under the curve over 24 hours using CGMS for breakfast, lunch, snack and dinner.
substrate oxidation | 3 hours post consumption
  Carbohydrate, fat and protein oxidation and respiratory quotient after consumption of low and high GI test foods are calculated for the 3 hours postprandial after breakfast, lunch and snack. These are calculated from the oxygen consumption, carbon dioxide production and nitrogen production. These sub-measurements are specified under: Other Pre-specified Outcomes: Oxygen consumption, carbon dioxide production, nitrogen production.
energy expenditure | 3 hours post consumption
  Energy expenditure after consumption of low and high GI test foods is calculated for the 3 hours postprandial after breakfast, lunch and snack. This is calculated from the oxygen consumption and carbon dioxide production. These sub-measurements are specified under: Other Pre-specified Outcomes: Oxygen consumption, carbon dioxide production.

OTHER OUTCOMES:
Oxygen consumption | 3 hours post consumption
  Oxygen consumption after consumption of low and high GI test foods measured 3 hours postprandial using indirect calorimetry in a whole body calorimeter. This is done over 10 hours in the whole body calorimeter measured for breakfast, lunch and snack only.
carbon dioxide production | 3 hours post consumption
  Carbon dioxide production after consumption of low and high GI test foods measured 3 hours postprandial using indirect calorimetry in a whole body calorimeter. This is done over 10 hours in the whole body calorimeter measured for breakfast, lunch and snack only.
Nitrogen production | 10 hours
  Nitrogen production during 10 hours in the whole body calorimeter is measured from all urine collected during the stay in the whole body calorimeter when consuming low and high GI test foods

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No